CLINICAL TRIAL: NCT03261310
Title: Use of IV Acetaminophen in the Treatment of Post Operative Pain in Patients Undergoing Craniotomy and Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dimitar Dentchev, Staff Anesthesiologist, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 386486-1
Record Dates: First submitted 2014-04-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Pain
Keywords: acetaminophen; pain; laminectomy; craniotomy
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acetaminophen & Craniotomy (Experimental): Drug: Acetaminophen 1000mg administered intravenously during craniotomy
  Interventions: Drug: Acetaminophen or Placebo
- Placebo & Craniotomy (Placebo Comparator): Placebo administered intravenously during craniotomy.
  Interventions: Drug: Acetaminophen or Placebo
- Acetaminophen & Laminectomy (Experimental): Acetaminophen 1000mg administered intravenously during laminectomy.
  Interventions: Drug: Acetaminophen or Placebo
- Placebo & Laminectomy (Placebo Comparator): Placebo administered during laminectomy.
  Interventions: Drug: Acetaminophen or Placebo

INTERVENTIONS:
Drug: Acetaminophen or Placebo — Study subject will receive either 1000mg of acetaminophen in 100ml own diluent, or 100ml of saline during their intra-operative period and an order will be placed in their chart/Essentris order for "No acetaminophen for 6 hours post operatively".

SUMMARY:
The purpose of this study is to investigate the effectiveness of intravenous acetaminophen (Tylenol) for post operative pain control in patients undergoing craniotomies (brain surgery) and spine surgery. Studies have shown that intravenous acetaminophen is useful for post operative pain control in some operations but there have not been studies to evaluate the use of acetaminophen in craniotomies or spine surgery.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effectiveness of intravenous acetaminophen (Tylenol) for post operative pain control in patients undergoing craniotomies (brain surgery) and spine surgery. Studies have shown that intravenous acetaminophen is useful for post operative pain control in some operations but there have not been studies to evaluate the use of acetaminophen in craniotomies or spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* undergoing non-emergent craniotomy or single level lumbar laminectomy
* must be able to rate pain on a 0-10 scale post-operatively

Exclusion Criteria:

* history of liver disease
* allergy to acetaminophen
* age less than 18 years
* renal failure with creatinine clearance less than 30
* pregnancy
* altered mentation with inability to report pain score
* patients who have received acetaminophen within 6 hours of surgery
* patients in which a neuraxial technique has been performed for surgery
* prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | 1hour -6 hours
  Primary outcomes will be measured pain scores at post-operative timepoints (1, 2, 4 and 6 hours), and the calculated percent change from baseline (1 hr post-op) for each of the follow-up pain scores (2, 4, 6 hours).

SECONDARY OUTCOMES:
Opioid administration | 1 hour-6 hours
  Secondary outcome will be a comparison of morphine equivalent dosages of opioid administered during the same periods between the treatment and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar Dentchev, MD, Principal Investigator — BAMC; Betsy Murray, MD, Study Chair — BAMC; Robert Vietor, MD, Study Chair — BAMC; Jonathan Deeth, MD, Study Chair — BAMC; Daniel Stypula, DO, Study Chair — BAMC
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided